CLINICAL TRIAL: NCT02071784
Title: Etude Comparative en Imagerie Par résonnance magnétique et Par Enregistrement électroencéphalographique du Couplage Neurovasculaire Dans l'Angiopathie Cadasil
Brief Title: Imaging Study of Neurovascular Coupling in Cerebral Autosomal Dominant Arteriopathy With Subcortical Infarcts and Leukoencephalopathy (CADASIL)
Acronym: MACOUPLING-CAD
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C13-62; 2014-A00200-47 (Registry Identifier: IDRCB)
Record Dates: First submitted 2014-02-24; First posted 2014-02-26 (Estimated); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: CADASIL
MeSH Terms: conditions — CADASIL

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to investigate using fMRI methods, EEG and dedicated mathematical models, the potential alterations of neurovascular coupling in CADASIL.

DETAILED DESCRIPTION:
Comparison study of parameters derived from mathematical models of neurovascular coupling and obtained using fMRI (Bold signal, ASL and EEG).

ELIGIBILITY:
Inclusion Criteria:

* CADASIL group: typical NOTCH3 mutation, age less than 60 years, rankin score at 0-1, active social insurance

Exclusion Criteria:

* MRI contra-indications and use of any treatment known to interfere with neurovascular coupling, pregnancy, lack of informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: CADASIL patients compared to age-matched controls (two groups)
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-07-08 (Actual); Primary Completion 2016-10-24 (Actual); Study Completion 2016-10-24 (Actual)

PRIMARY OUTCOMES:
model-derived parameters of neurovascular coupling | one time point

CONTACTS AND LOCATIONS:
Overall Officials: Hugues Chabriat, MD PhD, Principal Investigator — INSERM and APHP
Locations (1):
- CENIR, Hopital Pitié Salpetriere, Paris, France